CLINICAL TRIAL: NCT06685549
Title: The Relationship Between Isolated Head Trauma During Pregnancy and Preterm Birth
Acronym: PB
Status: Completed | Type: Observational
Sponsor: Sanliurfa Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Alev Esercan, Dr., Sanliurfa Education and Research Hospital
Other Study IDs: SEAH
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Superficial Injuries Involving Head With Neck
Keywords: cervical dilatation; head trauma; preterm birth; placental abruption; vaginal bleeding
MeSH Terms: conditions — Craniocerebral Trauma; Premature Birth; Abruptio Placentae; Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant patients after first trimester without any complaint: Patients with a similar age and gestational age, who were not exposed to any trauma, who had no health problems, and who applied to the outpatient clinic for follow-up were randomized with a computer program and formed a control group. The birth week, birth weight, type of birth, and admission to the neonatal intensive care unit of the control group were evaluated.
- isolated head trauma and pregnancy group: The criteria for inclusion in the study were as follows: all of the pregnant women over 18 years of age with isolated head trauma (closed blunt trauma) who were evaluated with neurosurgical consultation or computed tomography/magnetic resonance (CT/MRI) and whose birth records are available at our hospital.

SUMMARY:
Pregnant patients who presented to the Emergency Department of Şanlıurfa Training and Research Hospital with isolated head trauma due between January 2018 and January 2024 were included in the study and followed up with until the time of pregnancy termination.

DETAILED DESCRIPTION:
The criteria for inclusion in the study were as follows: all of the pregnant women over 18 years of age with isolated head trauma (closed blunt trauma) who were evaluated with neurosurgical consultation or computed tomography/magnetic resonance (CT/MRI) and whose birth records are available at our hospital.

The exclusion criteria included patients with previous premature birth, pregnancies in the first trimester, pregnancies with assisted reproductive techniques, multiple pregnancy, the threat of preterm labor or abortus imminens in the current pregnancy, maternal or fetal life-threatening situations that may cause termination of the pregnancy, cervical insufficiency, short cervix or history of conization, asymptomatic bacteriuria, periodontal disease, and smoking and substance use. Patients who had trauma to the other parts of the body or placental abruption were also excluded. Additionally, the study did not include those with missing hospital records regarding birth and pregnancy follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All of the pregnant women over 18 years of age with isolated head trauma (closed blunt trauma) who were evaluated with neurosurgical consultation or computed tomography/magnetic resonance (CT/MRI) and whose birth records are available at our hospital.

Exclusion Criteria:

Patients with previous premature birth, Pregnancies in the first trimester, Pregnancies with assisted reproductive techniques, Multiple pregnancy, The threat of preterm labor or abortus imminens in the current pregnancy, Maternal or fetal life-threatening situations that may cause termination of the pregnancy, Cervical insufficiency, Short cervix or history of conization, Diagnosis of asymptomatic bacteriuria, Diagnosis of periodontal disease, Smoking and substance use. Patients who had trauma to the other parts of the body or placental abruption Missing hospital records regarding birth and pregnancy follow-up.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant patients who presented to the Emergency Department of Şanlıurfa Training and Research Hospital with isolated head trauma due between January 2018 and January 2024 were included in the study and followed up with until the time of pregnancy termination.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
results of isolated head trauma | following maximum time for 6 months, until each pregnant's birth
  CT/MRI result of the patients' head trauma, whether they had surgery on the brain after the trauma, ward or intensive care hospitalizations
birth results | following maximum time for 6 months, until each pregnant's birth
  gestational week at birth
preterm birth results | following maximum time for 6 months, until each pregnant's birth
  whether preterm birth occurs, the baby's delivery method and weight

CONTACTS AND LOCATIONS:
Overall Officials: Alev Esercan, Assoc. Prof., Study Director — Sanliurfa Education and Research Hospital
Locations (1):
- Sanliurfa Training and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.uptodate.com/contents/spontaneous-preterm-birth-overview-of-risk-factors-and-prognosis?search=preterm%20birth&source=search_result&selectedTitle=1%7E150&usage_type=default&display_rank=1.